CLINICAL TRIAL: NCT04360356
Title: Clinical Trial Evaluating Safety and Efficacy of Ivermectin and Nitazoxanide Combination as Adjuvant Therapy in COVID-19 Newly Diagnosed Egyptian Patients: A Tanta University Hope
Brief Title: Ivermectin and Nitazoxanide Combination Therapy for COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kamal Mohammed Okasha, Vice-President of Postgraduate Studies and Research Affairs, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVR/NTZ
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Ivermectin; Nitazoxanide; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; nitazoxanide; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study will be a double blind randomized controlled parallel study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin plus Nitazoxanide (Experimental): Ivermectin 200 mcg/kg once orally on empty stomach plus Nitazoxanide 500 mg twice daily orally with meal for 6 days
  Interventions: Combination Product: Ivermectin plus Nitazoxanide
- Standard care (Active Comparator): Oxygen via ventilators
  Interventions: Other: Standard Care

INTERVENTIONS:
Combination Product: Ivermectin plus Nitazoxanide — Ivermectin 200 mcg/kg once orally on empty stomach plus Nitazoxanide 500 mg twice daily orally with meal for 6 days
  Arms: Ivermectin plus Nitazoxanide
Other: Standard Care — Oxygen via Ventilators
  Arms: Standard care

SUMMARY:
Research Background and Rationale

In December 2019, a new infectious respiratory disease emerged in Wuhan, Hubei province, China. An initial cluster of infections was linked to Huanan seafood market, potentially due to animal contact. Subsequently, human-to-human transmission occurred and the disease, now termed coronavirus disease 19 (COVID-19) rapidly spread within China and all over the world. A novel coronavirus, SARS-coronavirus 2 (SARS-CoV-2), which is closely related to SARS-CoV, was detected in patients and is believed to be the etiologic agent of the new lung disease. The causative agent of the current COVID-19 pandemic, SARS-CoV-2, is a single stranded positive sense RNA virus that is closely related to severe acute respiratory syndrome coronavirus (SARS-CoV).

DETAILED DESCRIPTION:
Selected Drugs

Ivermectin has anti-parasitic effect along with anti-viral activity against a broad range of viruses in vitro. Ivermectin was identified as an inhibitor of interaction between the human immunodeficiency virus-1 (HIV-1) integrase protein (IN) and the importin (IMP) α/β1 heterodimer responsible for IN nuclear import. Ivermectin has since been confirmed to inhibit HIV-1 replication. Importantly, Ivermectin has been demonstrated to limit infection by RNA viruses such as West Nile Virus and influenza. This broad-spectrum activity is believed to be due to the reliance by many different RNA viruses on IMPα/β1 during infection. Ivermectin has similarly been shown to be effective against the DNA virus pseudorabies virus (PRV) both in vitro and in vivo. Finally, Ivermectin was the focus of a phase III clinical trial in Thailand against DENV infection, in which a single daily oral dose was observed to be safe and resulted in a significant reduction in serum levels of viral NS1 protein, but no change in viremia or clinical benefit was observed.

The causative agent of the current COVID-19 pandemic, SARS-CoV-2, is a single stranded positive sense RNA virus that is closely related to severe acute respiratory syndrome coronavirus (SARS-CoV). Studies on SARS-CoV proteins have revealed a potential role for IMPα/β1 during infection in signal-dependent nucleocytoplasmic shutting of the SARS-CoV nucleocapsid protein that may impact host cell division. In addition, the SARS-CoV accessory protein ORF6 has been shown to antagonize the antiviral activity of the STAT1 transcription factor by sequestering IMPα/β1 on the rough ER/Golgi membrane.

Taken together, these reports suggested that Ivermectin's nuclear transport inhibitory activity may be effective against SARS-CoV-2. Interestingly, it has been postulated that the FDA-approved drug Ivermectin inhibits the replication of SARS-CoV-2 in vitro whereas a single treatment was able to provoke approximately 5000-fold reduction in viral load within 48h. Ivermectin has an established safety profile for human use. Recent reviews and meta-analysis indicate that high dose Ivermectin has comparable safety as the standard low-dose treatment, although there is not enough evidence to make conclusion about the safety profile in pregnancy. In clinical setting, Ivermectin was the focus of a phase III clinical trial on patients with dengue viral infection in Thailand, in which a single daily dose (200 - 400 µg/kg once daily for 2 days in one arm and 200-400 µg/kg once daily for 3 days in the other arm) was found to be safe but did not produce any clinical benefit. In previous clinical study, one dose of Ivermectin 200 μg/kg or four doses of Ivermectin 200 μg/kg (given on days 1, 2, 15, and 16) for the treatment of non-disseminated strongyloidiasis were implicated. The author proposed that, multiple doses of Ivermectin did not show higher efficacy and was tolerated less than a single dose. A single dose should, therefore, be preferred for the treatment of non-disseminated strongyloidiasis.

Nitazoxanide is originally developed as an antiprotozoal agent and has a broad-spectrum antiviral activity undergoing development for the treatment of influenza and other viral respiratory infections. In addition to its antiviral activity, Nitazoxanide inhibits the production of pro-inflammatory cytokines TNFα, IL-2, IL-4, IL-5, IL-6, IL-8 and IL-10 in peripheral blood mononuclear cells. Nitazoxanide could improve outcomes in patients infected with MERS-CoV by suppressing overproduction of pro-inflammatory cytokines, including IL-6. Nitazoxanide has been tested in clinical setting for the treatment of acute uncomplicated influenza, where the subjects received either 600 or 300 mg of Nitazoxanide or placebo orally twice daily for five days and were followed for 28 days. Subjects who received Nitazoxanide 600 mg twice daily experienced shorter times to alleviation of symptoms compared with subjects who received 300 mg Nitazoxanide twice daily, which in turn, was shorter than placebo.

According to the National Health Commission of the People's Republic of China, there is lack of effective antiviral therapy against COVID-19. Nearly all patients who suffered from COVID-19-associated pneumonia accepted oxygen therapy and WHO recommended extracorporeal membrane oxygenation (ECMO) to patients with refractory hypoxemia. Rescue treatment with convalescent plasma and immunoglobulin G are delivered to some critical cases according to their condition.

The rationale of the use of Ivermectin and Nitazoxanide combination for treatment of COVID-19 infected patients is based on the antiviral and anti-inflammatory activity of the selected drugs. Since the two drugs exhibit different modes of action, it would be of value in containing the viral infection through targeting different sites in the pathophysiology of the disease.

Diagnostic criteria

The viral research institution in China has conducted preliminary identification of the SARS-CoV-2 through the classical Koch's postulates and observing its morphology through electron microscopy. So far, the golden clinical diagnosis method of COVID-19 is nucleic acid detection in the nasal and throat swab sampling or other respiratory tract samplings by real-time PCR and further confirmation by next-generation sequencing.

Common Side Effects of Ivermectin

* Itching and rash
* Swelling
* Headache
* Joint pain
* Pink eye, inflammation of the eyes or discomfort
* Dizziness and drop in blood pressure upon standing
* Racing heart beat
* Changes in liver function tests
* Serious Side Effects of Ivermectin (Generally with Ivermectin tablets)
* Severe skin reactions
* Seizures
* Asthma flare-up
* Changes in vision
* Sudden drop in blood pressure
* Dizziness upon standing
* Liver dysfunction
* Bleeding

Drug interactions of Ivermectin

1. Warfarin and Coumarin Ivermectin may decrease the anticoagulant activities of warfarin and 4-hydroxycoumarin
2. Albendazole The metabolism of Albendazole can be increased when combined with Ivermectin
3. Doxycyline

Additive pharmacodynamic effect

* Contraindication of Ivermectin
* Abnormal liver function tests
* Allergies towards Ivermectin
* Side effects of Nitazoxanide
* The most common adverse effects are GIT as nausea and occasional stomach cramps with mild diarrhea, reduced appetite and vomiting. Nervous system side effects as headache, dizziness, somnolence, insomnia, tremor, and hypesthesia have been reported in less than 1% of the patients.

Contraindications of Nitazoxanide

* There are no data on the excretion of Nitazoxanide into human milk. The manufacturer recommends that caution should be used when administering Nitazoxanide to nursing women.

Interactions of Nitazoxanide

* Tizoxanide (the active metabolite of Nitazoxanide) is highly bound to plasma protein (> 99.9%). Therefore, it is necessary to monitor for adverse reactions when administering Nitazoxanide concurrently with other highly plasma protein-bound drugs with narrow therapeutic indices, as competition for binding sites may occur (e.g., warfarin).

Warning

* Nitazoxanide should be used with caution in patients with significant renal and hepatic impairment.

Research Objectives

The pandemic disease COVID-19 is particularly of major importance in Egypt where a heavy population lives. There is an acute need for comprehensive, continuous, and cost-effective health care delivery for infected people. Early detection and strategies for prevention of progression of COVID-19 would make a major difference for these patients and would also be economically beneficial for a resource-constrained country.

This research proposal was employed as a practical strategy for providing a suitable drug combination for possible treatment of COVID-19 infected patients. This drug combination may help to prevent the progression of respiratory complications. This can be achieved through different goals as follows:

1. Screening of different drugs related to different pharmacological classes depending on its possible activity against COVID-19 virus.
2. Providing cost-effective and easy-to-implement treatment strategy for infected patients and/or patients with high risk of developing respiratory failure.
3. Finally, this clinical strategy remains an important goal in improving Egyptian health state which can save people life and save a lot of money.

Scope of Work

The scope of work will be conducted through

1. Use of new drug combination of Ivermectin and Nitazoxanide for treatment of COVID-19 infected people. Since the two drugs exhibit different modes of action, it would be of value in containing the viral infection through targeting different sites in the pathophysiology of the disease.
2. Evaluation of the effect of new drug combination on the symptomatic treatment of COVID-19 patients according to WHO (Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected) interim guidance published at 13 March 2020.
3. Investigating the impact of new drug combination on the prevention of severe compilations such as acute respiratory distress syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

* Adult symptomatic patients (18-65 years old), both sexes, and PCR positive in nasopharyngeal sample at admission.

Exclusion Criteria:

* Abnormal liver function (ALT, AST), chronic kidney disease or dialysis (CrCl< 30 ml/min), immunocompromised patients taking medication upon screening, subjects on warfarin or dicumarol therapy and those with comorbid condition like hypertension, hypotension, cardiovascular disease, diabetes mellitus, asthma, COPD, seizures, coagulation disorder and malignancy.
* Patients will be also excluded if they had a known allergy to Ivermectin and/or Nitazoxanide, and those with contraindication towards the study medication.
* Pregnant women or women who are breastfeeding will be also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with COVID-19-negative PCR | within 10 days
  COVID-19 PCR analysis

SECONDARY OUTCOMES:
Number of patients with improved respiratory rate | within 30 days
  improved breaths per minute for the patients
Number of patients with improved PaO2 | within 30 days
  Change in PaO2 in mmHg of the patients
Number of patients with normalized Serum IL6 | within 30 days
  Serum IL6 in pg/mL of the patients
Number of patients with normalized Serum TNFα | within 30 days
  Serum TNFα in pg/mL of the patients
Number of patients with normalized Serum iron | within 30 days
  Serum iron in microgram/dL of the patients
Number of patients with normalized Serum ferritin | within 30 days
  Serum ferritinin microgram/L of the patients
Number of patients with normalized International normalized ratio "INR" for prothrombin time | within 30 days
  International normalized ratio "INR" for prothrombin time of 2
Number of patients with normalized complete blood count "CBC" | within 30 days
  CBC for lymphocyte count in cells/microliter
The Mortality rate among treated patients | within 30 days
  Mortality rate [number of dead patients/total number of treated patients]

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Okasha, Md, PhD, Principal Investigator — Tanta University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Wagstaff KM, Rawlinson SM, Hearps AC, Jans DA. An AlphaScreen(R)-based assay for high-throughput screening for specific inhibitors of nuclear import. J Biomol Screen. 2011 Feb;16(2):192-200. doi: 10.1177/1087057110390360. PMID 21297106
- [Background] Gotz V, Magar L, Dornfeld D, Giese S, Pohlmann A, Hoper D, Kong BW, Jans DA, Beer M, Haller O, Schwemmle M. Influenza A viruses escape from MxA restriction at the expense of efficient nuclear vRNP import. Sci Rep. 2016 Mar 18;6:23138. doi: 10.1038/srep23138. PMID 26988202
- [Background] Jans DA, Martin AJ, Wagstaff KM. Inhibitors of nuclear transport. Curr Opin Cell Biol. 2019 Jun;58:50-60. doi: 10.1016/j.ceb.2019.01.001. Epub 2019 Feb 28. PMID 30826604
- [Background] Lv C, Liu W, Wang B, Dang R, Qiu L, Ren J, Yan C, Yang Z, Wang X. Ivermectin inhibits DNA polymerase UL42 of pseudorabies virus entrance into the nucleus and proliferation of the virus in vitro and vivo. Antiviral Res. 2018 Nov;159:55-62. doi: 10.1016/j.antiviral.2018.09.010. Epub 2018 Sep 26. PMID 30266338
- [Background] Wulan WN, Heydet D, Walker EJ, Gahan ME, Ghildyal R. Nucleocytoplasmic transport of nucleocapsid proteins of enveloped RNA viruses. Front Microbiol. 2015 Jun 2;6:553. doi: 10.3389/fmicb.2015.00553. eCollection 2015. PMID 26082769
- [Background] Wurm T, Chen H, Hodgson T, Britton P, Brooks G, Hiscox JA. Localization to the nucleolus is a common feature of coronavirus nucleoproteins, and the protein may disrupt host cell division. J Virol. 2001 Oct;75(19):9345-56. doi: 10.1128/JVI.75.19.9345-9356.2001. PMID 11533198
- [Background] Frieman M, Yount B, Heise M, Kopecky-Bromberg SA, Palese P, Baric RS. Severe acute respiratory syndrome coronavirus ORF6 antagonizes STAT1 function by sequestering nuclear import factors on the rough endoplasmic reticulum/Golgi membrane. J Virol. 2007 Sep;81(18):9812-24. doi: 10.1128/JVI.01012-07. Epub 2007 Jun 27. PMID 17596301
- [Background] Navarro M, Camprubi D, Requena-Mendez A, Buonfrate D, Giorli G, Kamgno J, Gardon J, Boussinesq M, Munoz J, Krolewiecki A. Safety of high-dose ivermectin: a systematic review and meta-analysis. J Antimicrob Chemother. 2020 Apr 1;75(4):827-834. doi: 10.1093/jac/dkz524. PMID 31960060
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Hong SK, Kim HJ, Song CS, Choi IS, Lee JB, Park SY. Nitazoxanide suppresses IL-6 production in LPS-stimulated mouse macrophages and TG-injected mice. Int Immunopharmacol. 2012 May;13(1):23-7. doi: 10.1016/j.intimp.2012.03.002. Epub 2012 Mar 17. PMID 22430099
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516